CLINICAL TRIAL: NCT04592354
Title: Anhydrous Enol-Oxaloacetate (AEO) on Improving Fatigue in Post-COVID-19 Survivors
Acronym: AEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Terra Biological LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-AEO-2020 Post Covid Fatigue
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Treatment of Fatigue After Resolution of COVID-19 Infection

STUDY DESIGN:
Intervention Model Description: Double Blinded placebo controlled comparison study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded active and placebo groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxaloacetate Therapeutic Arm (Active Comparator): * Anhydrous Enol-Oxaloacetate
  * A 500 mg oxaloacetate capsule taken by mouth twice a day
  * Planned study duration is 6 weeks with an interim assessment at the end of 2 weeks and final assessment at 6 weeks
  Interventions: Dietary Supplement: Oxaloacetate Medical Food/Dietary Supplement
- Placebo Arm (Placebo Comparator): * Rice Flour
  * A 500 mg rice flour capsule taken by mouth twice a day
  Interventions: Dietary Supplement: Oxaloacetate Medical Food/Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Oxaloacetate Medical Food/Dietary Supplement — 500 mg Anhydrous Enol-Oxaloacetate BID

SUMMARY:
We will conduct a double arm, randomized, double-blinded placebo controlled trial of oxaloacetate for treatment of fatigue in women with a history of COVID-19 infection, resolution of the infection, and remaining fatigue that interfere with everyday activities, based on use of a standardized questionnaire to screen for impairment.

Participants will receive a 6-week supply of the active or placebo and will be asked to take one capsule twice a day with water and food. They will be contacted weekly for two weeks by the study coordinator to assess for any side effects or difficulty taking the medication. They will be asked to again to complete the standardized questionnaire to screen for impairment after 2 weeks, and again at the end of the study at 6 weeks. Finally, any adverse reactions and symptoms will be evaluated once again four weeks later to ensure that any symptoms that may have been present during treatment have resolved.

DETAILED DESCRIPTION:
We will conduct a double arm, randomized, double-blinded placebo controlled trial of oxaloacetate for treatment of fatigue in women with a history of COVID-19 infection, resolution of the infection, and remaining fatigue that interfere with everyday activities, based on use of a standardized questionnaire to screen for impairment. Women will be recruited from a variety of settings including clinics affiliated with our existing doctor base, outreach through social media and notification of community organizations that serve this patient population. The study will take place at the residences of the participants, being performed virtually after receipt of informed consent paperwork, COVID-19 positive test data, and COVID -19 negative resolution data by us, and by receipt of the test product by the participant. Efforts will be made to conduct as much of this trial virtually as possible due to the Covid-19 pandemic. Women who could potentially be pregnant will undergo pregnancy testing and determination of menopausal status, if appropriate. Participants will complete baseline questionnaires that assess fatigue and depressive symptoms.

Subsequently, the participants will receive a 6-week supply of the active or placebo and will be asked to take one capsule twice a day with water and food. They will be contacted weekly for two weeks by the study coordinator to assess for any side effects or difficulty taking the medication. They will be asked to again to complete the standardized questionnaire to screen for impairment after 2 weeks, and again at the end of the study at 6 weeks. Finally, any adverse reactions and symptoms will be evaluated once again four weeks later to ensure that any symptoms that may have been present during treatment have resolved.

ELIGIBILITY:
Inclusion Criteria:

* 4.1.1 Women with an initial infection diagnosis COVID-19 that has been resolved, as measured by rRT PCR, who are at least 2 months after proven viral resolution.
* 4.1.2 No evidence of active/recurrent COVID-19 or other serious chronic illness.
* 4.1.3 Have significant fatigue complaints, defined as a bimodal score of 4 or greater on the Fatigue Questionnaire.
* 4.1.4 Is geographically accessible, or can fill out forms virtually, and able to participate in a study of 6-10 weeks duration.
* 4.1.5 Age >18 years and less than 65.
* 4.1.6 Ability to complete evaluation surveys in English.
* 4.1.7 The effects of oxaloacetate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (barrier method of birth control; IUD; abstinence) prior to study entry and for the duration of study participation. Women of any age who have had their ovaries and/or uterus removed will not be at risk for pregnancy and will not require contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

  * Menopausal status will be established as follows: Women who are 55 years or older and who are not menstruating will be considered postmenopausal and not at risk for pregnancy. Women who are less than 55 years old who are menstruating will be considered premenopausal and will require contraception. Women who are less than 55 years with an intact uterus and ovaries who are not menstruating and have not had a menstrual period within the past 2 years will have an FSH and estradiol measured. If the values are in postmenopausal range the woman will be considered postmenopausal and she will not be considered at risk for pregnancy.
* 4.1.8 Ability to understand and the willingness to sign a written informed consent document.
* 4.1.9 No diagnosis of Clinical Depression
* 4.1.10 Is not taking an oxaloacetate supplement.

Exclusion Criteria:

* 4.2.1 Has another serious or chronic medical or psychiatric condition that contributes to substantial physical or emotional disability that would detract from participating in the planned study.
* 4.2.2 Taking chronic medications that would interfere with cognitive functioning such as medications for sleep, anxiety, narcotics for pain, use of illicit medical foods or cannabis.
* 4.2.3 Participants may not be receiving any other investigational agents.
* 4.2.4 History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaloacetate.
* 4.2.5 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection of Covid-19 or other virus, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* 4.2.6 Pregnant or breast-feeding women are excluded from this study because the safety of oxaloacetate in this setting is unknown. A pregnancy test will be performed on all women with an intact uterus and ovaries who are not determined to be postmenopausal, as described in section 4.1.7.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 6 weeks
  Evaluation of self-reported Fatigue with the Fatigue Questionnaire (FQ)

SECONDARY OUTCOMES:
Fatigue | 6 weeks
  Evaluation of self-reported Fatigue with the Fatigue Severity Scale (FSS)
Depression | 6 weeks
  Evaluation of self-reported depression with Beck's Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tully, Ph.D., Principal Investigator — Energy Medicine Research Institute
Locations (1):
- Energy Medicine research Institute, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the data so that it is available to other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after the conclusion of the study
Access Criteria: Unknown at this point.

REFERENCES:
- [Background] Rasa S, Nora-Krukle Z, Henning N, Eliassen E, Shikova E, Harrer T, Scheibenbogen C, Murovska M, Prusty BK; European Network on ME/CFS (EUROMENE). Chronic viral infections in myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). J Transl Med. 2018 Oct 1;16(1):268. doi: 10.1186/s12967-018-1644-y. PMID 30285773
- [Background] Lyons D, Frampton M, Naqvi S, Donohoe D, Adams G, Glynn K. Fallout from the COVID-19 pandemic - should we prepare for a tsunami of post viral depression? Ir J Psychol Med. 2020 Dec;37(4):295-300. doi: 10.1017/ipm.2020.40. Epub 2020 May 15. PMID 32408926
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Ettman CK, Abdalla SM, Cohen GH, Sampson L, Vivier PM, Galea S. Prevalence of Depression Symptoms in US Adults Before and During the COVID-19 Pandemic. JAMA Netw Open. 2020 Sep 1;3(9):e2019686. doi: 10.1001/jamanetworkopen.2020.19686. PMID 32876685
- [Background] Yamamoto HA, Mohanan PV. Effect of alpha-ketoglutarate and oxaloacetate on brain mitochondrial DNA damage and seizures induced by kainic acid in mice. Toxicol Lett. 2003 Jul 20;143(2):115-22. doi: 10.1016/s0378-4274(03)00114-0. PMID 12749815
- [Background] Campos F, Sobrino T, Ramos-Cabrer P, Castillo J. Oxaloacetate: a novel neuroprotective for acute ischemic stroke. Int J Biochem Cell Biol. 2012 Feb;44(2):262-5. doi: 10.1016/j.biocel.2011.11.003. Epub 2011 Nov 10. PMID 22085530
- [Background] Ruban A, Berkutzki T, Cooper I, Mohar B, Teichberg VI. Blood glutamate scavengers prolong the survival of rats and mice with brain-implanted gliomas. Invest New Drugs. 2012 Dec;30(6):2226-35. doi: 10.1007/s10637-012-9799-5. PMID 22392507
- [Background] Nagy D, Marosi M, Kis Z, Farkas T, Rakos G, Vecsei L, Teichberg VI, Toldi J. Oxaloacetate decreases the infarct size and attenuates the reduction in evoked responses after photothrombotic focal ischemia in the rat cortex. Cell Mol Neurobiol. 2009 Sep;29(6-7):827-35. doi: 10.1007/s10571-009-9364-8. Epub 2009 Mar 4. PMID 19259807
- [Background] Zlotnik A, Gurevich B, Tkachov S, Maoz I, Shapira Y, Teichberg VI. Brain neuroprotection by scavenging blood glutamate. Exp Neurol. 2007 Jan;203(1):213-20. doi: 10.1016/j.expneurol.2006.08.021. Epub 2006 Oct 2. PMID 17014847
- [Background] Nagy D, Knapp L, Marosi M, Farkas T, Kis Z, Vecsei L, Teichberg VI, Toldi J. Effects of blood glutamate scavenging on cortical evoked potentials. Cell Mol Neurobiol. 2010 Oct;30(7):1101-6. doi: 10.1007/s10571-010-9542-8. Epub 2010 Jul 6. PMID 20607387
- [Background] Swerdlow RH, Bothwell R, Hutfles L, Burns JM, Reed GA. Tolerability and pharmacokinetics of oxaloacetate 100 mg capsules in Alzheimer's subjects. BBA Clin. 2016 Mar 10;5:120-3. doi: 10.1016/j.bbacli.2016.03.005. eCollection 2016 Jun. PMID 27051598
- [Background] Vidoni ED, Choi IY, Lee P, Reed G, Zhang N, Pleen J, Mahnken JD, Clutton J, Becker A, Sherry E, Bothwell R, Anderson H, Harris RA, Brooks W, Wilkins HM, Mosconi L, Burns JM, Swerdlow RH. Safety and target engagement profile of two oxaloacetate doses in Alzheimer's patients. Alzheimers Dement. 2021 Jan;17(1):7-17. doi: 10.1002/alz.12156. Epub 2020 Jul 27. PMID 32715609
- [Background] Matsos A, Johnston IN. Chemotherapy-induced cognitive impairments: A systematic review of the animal literature. Neurosci Biobehav Rev. 2019 Jul;102:382-399. doi: 10.1016/j.neubiorev.2019.05.001. Epub 2019 May 4. PMID 31063740
- [Background] Dantzer R, Kelley KW. Twenty years of research on cytokine-induced sickness behavior. Brain Behav Immun. 2007 Feb;21(2):153-60. doi: 10.1016/j.bbi.2006.09.006. Epub 2006 Nov 7. PMID 17088043
- [Background] Haroon E, Miller AH, Sanacora G. Inflammation, Glutamate, and Glia: A Trio of Trouble in Mood Disorders. Neuropsychopharmacology. 2017 Jan;42(1):193-215. doi: 10.1038/npp.2016.199. Epub 2016 Sep 15. PMID 27629368
- [Background] Boyko M, Gruenbaum SE, Gruenbaum BF, Shapira Y, Zlotnik A. Brain to blood glutamate scavenging as a novel therapeutic modality: a review. J Neural Transm (Vienna). 2014 Aug;121(8):971-9. doi: 10.1007/s00702-014-1181-7. Epub 2014 Mar 13. PMID 24623040
- [Background] Missailidis D, Annesley SJ, Allan CY, Sanislav O, Lidbury BA, Lewis DP, Fisher PR. An Isolated Complex V Inefficiency and Dysregulated Mitochondrial Function in Immortalized Lymphocytes from ME/CFS Patients. Int J Mol Sci. 2020 Feb 6;21(3):1074. doi: 10.3390/ijms21031074. PMID 32041178
- [Background] Nilsson I, Palmer J, Apostolou E, Gottfries CG, Rizwan M, Dahle C, Rosen A. Metabolic Dysfunction in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Not Due to Anti-mitochondrial Antibodies. Front Med (Lausanne). 2020 Mar 31;7:108. doi: 10.3389/fmed.2020.00108. eCollection 2020. PMID 32296708
- [Background] Wilkins HM, Harris JL, Carl SM, E L, Lu J, Eva Selfridge J, Roy N, Hutfles L, Koppel S, Morris J, Burns JM, Michaelis ML, Michaelis EK, Brooks WM, Swerdlow RH. Oxaloacetate activates brain mitochondrial biogenesis, enhances the insulin pathway, reduces inflammation and stimulates neurogenesis. Hum Mol Genet. 2014 Dec 15;23(24):6528-41. doi: 10.1093/hmg/ddu371. Epub 2014 Jul 15. PMID 25027327
- [Background] Katz JN, Chang LC, Sangha O, Fossel AH, Bates DW. Can comorbidity be measured by questionnaire rather than medical record review? Med Care. 1996 Jan;34(1):73-84. doi: 10.1097/00005650-199601000-00006. PMID 8551813
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Sloan JA, Loprinzi CL, Novotny PJ, Barton DL, Lavasseur BI, Windschitl H. Methodologic lessons learned from hot flash studies. J Clin Oncol. 2001 Dec 1;19(23):4280-90. doi: 10.1200/JCO.2001.19.23.4280. PMID 11731510
- [Derived] Cash A, Kaufman DL. Oxaloacetate Treatment For Mental And Physical Fatigue In Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and Long-COVID fatigue patients: a non-randomized controlled clinical trial. J Transl Med. 2022 Jun 28;20(1):295. doi: 10.1186/s12967-022-03488-3. PMID 35764955